CLINICAL TRIAL: NCT02644824
Title: Biventricular Pacing in Children With Wide QRS After Surgery for Congenital Heart Disease
Brief Title: Biventricular Pacing in Children With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Friedberg, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000032246
Record Dates: First submitted 2015-05-26; First posted 2016-01-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: Congenital Heart Disease (CHD); Cardiopulmonary Bypass (CPB); Cardiac Index; Hemodynamics; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biventricular Pacing (BiVp) (Experimental): Consented infants with wide QRS randomized to receive standard of care and BiVp.
  Interventions: Device: Biventricular Pacing (BiVp)
- Control (wide QRS) (No Intervention): Consented infants with wide QRS randomized to receive standard of care alone.
- Control (narrow QRS) (No Intervention): This is an observation control group. Consented infants with narrow QRS will enter control group 2 without randomization.

INTERVENTIONS:
Device: Biventricular Pacing (BiVp) — BiVp shortens QRS duration and synchronizes ventricular contraction; thereby decreasing wall stress and increasing CI and BP. In contrast to inotropes, BiVp does not increase myocardial VO2. Resynchronizing myocardial contraction normalizes glucose metabolism, myocardial perfusion and distribution of proteins essential to myocardial contraction and relaxation such as calcium-handling phospholamban. Overall, BiVp improves pump function, increases CI, improves myocardial perfusion and reduces VO2, improving hemodynamics.
  Arms: Biventricular Pacing (BiVp)

SUMMARY:
Surgery with cardiopulmonary bypass (CPB) for congenital heart disease (CHD) causes low cardiac index (CI). With the increasing success of surgery for CHD, mortality has decreased and emphasis has shifted to post-operative morbidity and recovery. Children with CHD undergoing surgery with CPB can experience well-characterized post-operative cardiac dysfunction. When severe, patients can develop clinically important low cardiac output syndrome (LCOS) and hemodynamic instability. Management of LCOS and hemodynamic compromise is primarily accomplished via intravenous durgs like milrinone, dopamine or dobutamine, which affect the strength of the heart's muscular contractions. These are used to maintain adequate blood pressure (BP) and CI. However, inotropic agents are potentially detrimental to myocardial function and may increase risk for post-operative arrhythmia and impair post-operative recovery by increasing oxygen demand and myocardial oxygen consumption (VO2). In combination with the increased VO2 associated with CPB-induced systemic inflammatory response patients can develop a critical mismatch between oxygen supply and demand, essentially the definition of LCOS. Therefore, therapies that improve CI and hemodynamic stability without increased VO2 are beneficial. This study will test whether BiVp, a specialized yet simple pacing technique, can improve post-operative CI and recovery in infants with electro-mechanical dyssynchrony (EMD) after CHD surgery. This study hypothesizes that Continuous BiVp increases the mean change in CI from baseline to 48 hours in infants with EMD following CHD surgery compared to standard care alone.

DETAILED DESCRIPTION:
Research Design: Pilot-study for a large prospective, randomized, single-blinded, clinical trial.

This study is a parallel-arm, randomized, single-blinded clinical trial based on a hemodynamic outcome that will inform a subsequent larger randomized trial based on clinical outcomes.

Main research question: Does continuous BiVp for up to 48 hours in infants with EMD after CHD surgery increase CI as measured every 1-3 hours by the Fick method using an AMIS2000 mass spectrometer for VO2 measurement? Primary Hypothesis: Continuous BiVp increases the mean change in CI from baseline to 48 hours in infants with EMD following CHD surgery compared to standard care alone.

Primary objective: The primary objective of this pilot study is to provide physiologic proof of principle data by testing the hypothesis that continuous BiVp increases the mean change in CI from baseline to 48 hours in infants with EMD following CHD surgery. Although this is suggested by our preliminary data, the number of infants with wide QRS was small and statistically underpowered. The current study will expand the target population and provide preliminary data for sample size calculation and outcome measures for a subsequent, larger, clinical trial based on clinical outcomes such as duration of mechanical ventilation, length of ICU stay and vasoactive-inotropic score.

Secondary Hypotheses:

1. BiVp reduces the maximum vasoactive-inotropic score over the 1st 48 hours after CHD surgery in infants with EMD compared to standard therapy.
2. BiVp improves end-organ perfusion: cerebral NIRS, serum lactate, kidney (time to negative fluid balance, creatinine clearance and neutrophil gelatinase-associated lipocalin (NGAL)), liver function (AST, ALT) and brain natiuretic peptide (BNP) in the 1st 48 hours in infants with EMD after CHD surgery compared to standard therapy.
3. BiVp reduces duration of mechanical ventilation in infants with EMD after CHD surgery.

Study population Screening: Potentially eligible patients will be screened by the study coordinator, Ms Rita Nobile, using the cardiovascular surgical schedule at SickKids. Consecutive patients will be enrolled to maximize representation of the target population. All screened patients will be registered in a screening log according to the CONSORT statement.60 Inclusion criteria-infants must meet all inclusion criteria to be enrolled: 1. Post-operative QRS duration ≥ 98th centile for age based on Davignon.61 2. 0-1 year of age undergoing biventricular repair of CHD under CPB. Based on a recent population undergoing CHD surgery over a 1-year period at SickKids, wthe investigators expect the following types of CHD to be included (Table 2, p.23): tetralogy of Fallot (40%), transposition of the great arteries (30%), complete atrioventricular septal defect (15%), interrupted aortic arch (4%), other (10%).

Exclusion criteria- Exclusion criteria will be assessed before and after surgery by the study coordinator and investigators. The presence of any criterion will exclude an infant from the study:

1. Extubation in operating room or expected extubation <12 hours after surgery. 2. Functionally univentricular heart disease (lack of septation into 2 ventricles each supporting pulmonary or systemic circulations). 3. Major extra-cardiac anomalies (expected to affect mechanical ventilation, ICU stay, 30-day mortality, expected to require intervention within 30-days, lethal genetic abn.(e.g. trisomy 13/18)). 4. Surgery without CPB or palliative surgery (e.g systemic-pulmonary shunt). 5. Weight <2.5 kg at time of surgery. 6. ECMO (at time of the ICU admission), infants expected to die or require ECMO within 12 hours after operation (judged by surgeon or ICU responsible physician); brain death within 12 hours after surgery (declared by ICU responsible physician). 7. Previous cardiac operation on CPB. 8. Junctional, atrial ectopic or ventricular tachycardia.

If BiVp (time zero in controls) has started and an arrhythmia precluding BiVp (listed above) or ECMO occurs ≤ 8 hrs after surgery, the patient will be excluded; if >8 hrs -analysis will be 'intention-to-treat'.

Study Groups: Following these inclusion/ exclusion criteria there will be 3 study groups:

1. Intervention group: Consented infants with wide QRS randomized to BiVp.
2. Control group 1: Consented infants with wide QRS randomized to the control group.
3. Control group 2 (observation group): Consented infants with narrow QRS will enter control group 2 without randomization. All study outcome measurements will be performed on this group. Enrolment, informed consent, randomization and definition of time zero: Informed signed consent will be obtained by the PIs and research coordinator from the infant's legal guardians prior to surgery. At surgery all consented patients will receive 3 temporary epicardial pacing leads: standard right atrial and RV leads, LV apical lead. On return to the intensive care unit, QRS width will be manually evaluated from an unpaced 12-lead ECG by Dr Stephenson, Friedberg or Schwartz. Children with prolonged QRS (≥98 centile61 by the longest QRS duration from any lead) (expected in ~48% of infants (Fig. 2, p.18) will be randomized in a 1:1 pacing: control ratio by computer-generated allocation (www.random.org) to receive either standard of care plus BiVp or to standard of care alone. Consented patients with QRS duration <98 centile will be allocated to the narrow QRS control group (control group 2). For the BiVp group time zero is defined by the start of pacing. For controls, time zero is 1 hour after arrival in the ICU (expected time BiVp will start in the intervention group).

ELIGIBILITY:
Inclusion Criteria:

* Infants 0-1 year with Congenital Heart Disease
* Patients with functionally univentricular heart disease
* Informed consent

Exclusion Criteria:

* Infants <2.5 kg at time of surgery
* Infants with biventricular heart disease
* Informed consent is not given

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac Index (CI) | Pre-operative, baseline, and every 24 hours during care up to 48 hours
  The overall mean change in CI from baseline (average of 1st 2 CI measurements) to study end (average of last 2 measurements) in BiVp vs. controls.

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation | From baseline to extubation at 48 hours
  Defined as fulfilling pre-defined, standard eligibility criteria for extubation: adequate gas exchange on an FiO2 of 30% or less, CPAP with pressure support of 10 cm H20, and no evidence of major pulmonary pathology on chest x-ray.
End Organ Perfusion | Pre-operative, baseline, and every 24 hours during care and up to 48 hours
  End organ perfusion will be assessed globally and in 3 major organ systems: 1) Kidneys 2) Brain 3) Liver. Globally, blood gases and serum lactate recovery will be used as indicators of organ perfusion.
QRS Duration | Pre-operative, baseline, and at study end of 48 hours
  QRS duration is a central measure of electro-mechanical dyssynchrony.QRS duration will be obtained pre-operatively, at baseline (arrival in intensive care unit before pacing) and every 24 hours with and without pacing. Computer generated QRS measurement may be more reliable than manual measurement when QRS is narrow, but all values will be confirmed manually from any lead on the 12-lead ECG.
Vasoactive-inotropic Score | Change from baseline of vasoactive-inotropic score to end of care and up to 48 hours
  Doses of vaso-active-inotropic agents at time of CI measurements will be recorded. A total vaso-active inotropic score will be calculated as the inotrope score + 10 x milrinone dose (µg/kg/min) + 10,000 x vasopressin dose (U/kg/min) + 100 x norepinephrine dose (µg/kg/min). The inotrope score is calculated as the dopamine dose (µg/kg/min) + dobutamine dose + 100 x epinephrine dose (µg/kg/min). Maximal vasoactive-inotropic score and change in vasoactive-inotropic score from baseline to study end will be assessed as secondary outcomes.
Mechanical Dyssynchrony | Pre-operative, baseline, and at study endat 48 hours
  Mechanical dyssynchrony will be investigated by echo before surgery, at baseline (in ICU before pacing) and at study end (before stopping pacing).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Friedberg, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada